CLINICAL TRIAL: NCT02040532
Title: Pilot Study to Assess Tolerability and Preliminary Efficacy of a Titrated Dose of Gabapentin up to 600mg Administered at Bedtime for Insomnia Symptoms and Nighttime Vasomotor Symptoms (VMS) in Peri- and Postmenopausal Women With VMS.
Brief Title: Gabapentin for Insomnia Symptoms and Nighttime Vasomotor Symptoms (VMS) in Peri- and Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lee S. Cohen, MD, Director, Center for Women's Mental Health, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013P002196; 5U01AG032700-05 (NIH)
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Menopause; Hot Flashes; Vasomotor Disturbance
MeSH Terms: conditions — Hot Flashes | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label gabapentin (Experimental): Dose titration of 100mg for 1 week, 300mg for 3 weeks, and 600mg for 3 weeks.
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — The study is a 7-week intervention study using open-label gabapentin at bedtime with a scheduled dose titration from 100-mg for one week, followed by 300-mg for 3 weeks, and then 600-mg for 3 weeks.
  Other Names: Neurontin

SUMMARY:
The broad goal of this study is to obtain pilot data to determine the tolerability and preliminary efficacy of the non-hormonal agent gabapentin for insomnia symptoms and nighttime vasomotor Symptoms (VMS) when open-label gabapentin is administered at low dose and only at night in peri- and postmenopausal women. We hypothesize that the majority of participants will be able to increase and tolerate treatment, and insomnia symptoms and the frequency of nighttime VMS will improve on low-dose gabapentin dosed at bedtime.

DETAILED DESCRIPTION:
Thirty-two peri- and postmenopausal women at the Boston sites (MGH and BWH) were enrolled into this open-label pilot study. The study was a 7-week intervention study using open-label gabapentin at bedtime with a scheduled dose titration from 100-mg for one week, followed by 300-mg for 3 weeks, and then 600-mg for 3 weeks. The intervention study followed a 3-week screening period to establish a stable baseline for insomnia symptoms and VMS and to determine the safety of administering gabapentin in study participants. Tolerability and treatment response (insomnia symptoms, nighttime VMS) were assessed systematically at each study visit. The dose titration schedule was followed in all participants unless there are dose-limiting toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 40-65 years
2. Postmenopausal or perimenopausal
3. Having bothersome hot flashes
4. Having some bothersome hot flashes during the night
5. Insomnia or problems sleeping
6. In general, good health
7. Signed informed consent

Exclusion Criteria:

1. Recent use of hormone therapy or hormonal contraceptives (with the exception of the Mirena IUD)
2. Recent use of any prescribed therapy that is taken specifically for hot flashes
3. Recent use of any over-the-counter or herbal therapies that are taken specifically for hot flashes
4. Recent use of any prescribed medications with known hot flash efficacy
5. Known hypersensitivity or contraindications (reasons not to take) to gabapentin
6. Not using a medically approved method of birth control, if sexually active and not 12 or more months since last menstrual period
7. Recent drug or alcohol abuse
8. Lifetime diagnosis of psychosis or bipolar disorder
9. Suicide attempt in the past 3 years or any current suicidal ideation
10. Current major depression (assessed during screening)
11. Pregnancy, intending pregnancy, or breast feeding
12. History of:

    1. Renal insufficiency or a kidney disorder
    2. Sleep disorder diagnosis of sleep apnea, restless legs syndrome, periodic limb movement disorder, or narcolepsy
13. Any unstable medical condition
14. Working a night/rotating shift
15. Abnormal screening blood tests
16. Current participation in another drug trial or intervention study
17. Inability or unwillingness to complete the study procedures

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee S Cohen, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ensrud KE, Joffe H, Guthrie KA, Larson JC, Reed SD, Newton KM, Sternfeld B, Lacroix AZ, Landis CA, Woods NF, Freeman EW. Effect of escitalopram on insomnia symptoms and subjective sleep quality in healthy perimenopausal and postmenopausal women with hot flashes: a randomized controlled trial. Menopause. 2012 Aug;19(8):848-55. doi: 10.1097/gme.0b013e3182476099. PMID 22433978
- [Background] Joffe H, Petrillo L, Viguera A, Koukopoulos A, Silver-Heilman K, Farrell A, Yu G, Silver M, Cohen LS. Eszopiclone improves insomnia and depressive and anxious symptoms in perimenopausal and postmenopausal women with hot flashes: a randomized, double-blinded, placebo-controlled crossover trial. Am J Obstet Gynecol. 2010 Feb;202(2):171.e1-171.e11. doi: 10.1016/j.ajog.2009.10.868. Epub 2009 Dec 24. PMID 20035910
- [Background] Soares CN, Joffe H, Rubens R, Caron J, Roth T, Cohen L. Eszopiclone in patients with insomnia during perimenopause and early postmenopause: a randomized controlled trial. Obstet Gynecol. 2006 Dec;108(6):1402-10. doi: 10.1097/01.AOG.0000245449.97365.97. PMID 17138773
- [Background] Yurcheshen ME, Guttuso T Jr, McDermott M, Holloway RG, Perlis M. Effects of gabapentin on sleep in menopausal women with hot flashes as measured by a Pittsburgh Sleep Quality Index factor scoring model. J Womens Health (Larchmt). 2009 Sep;18(9):1355-60. doi: 10.1089/jwh.2008.1257. PMID 19708803
- [Background] Butt DA, Lock M, Lewis JE, Ross S, Moineddin R. Gabapentin for the treatment of menopausal hot flashes: a randomized controlled trial. Menopause. 2008 Mar-Apr;15(2):310-8. doi: 10.1097/gme.0b013e3180dca175. PMID 17917611
- [Background] Pandya KJ, Morrow GR, Roscoe JA, Zhao H, Hickok JT, Pajon E, Sweeney TJ, Banerjee TK, Flynn PJ. Gabapentin for hot flashes in 420 women with breast cancer: a randomised double-blind placebo-controlled trial. Lancet. 2005 Sep 3-9;366(9488):818-24. doi: 10.1016/S0140-6736(05)67215-7. PMID 16139656
- [Background] Reddy SY, Warner H, Guttuso T Jr, Messing S, DiGrazio W, Thornburg L, Guzick DS. Gabapentin, estrogen, and placebo for treating hot flushes: a randomized controlled trial. Obstet Gynecol. 2006 Jul;108(1):41-8. doi: 10.1097/01.AOG.0000222383.43913.ed. PMID 16816054
- [Background] Aguirre W, Chedraui P, Mendoza J, Ruilova I. Gabapentin vs. low-dose transdermal estradiol for treating post-menopausal women with moderate to very severe hot flushes. Gynecol Endocrinol. 2010 May;26(5):333-7. doi: 10.3109/09513590903511539. PMID 20050764

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were recruited from the Boston area and enrolled at either the Massachusetts General Hospital Center for Women's Mental Health or the Brigham and Women's Hospital Women's Hormones and Aging Research Program.
Period: Overall Study
Arm/Group | Open-label Gabapentin
Started | 32
Received at Least One Dose of Medication | 26
Completed | 20
Not Completed | 12
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 4
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Gabapentin
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.31 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26
Highest Level of Education [Count of Participants; unit: Participants]
  Less than College Graduate | 18
  College Graduate/Baccalaureate Degree | 4
  Graduate Degree | 4
Employment [Count of Participants; unit: Participants]
  Employed Full-Time | 8
  Employed Part-Time | 6
  Retired or Unemployed | 8
  Disabled, Unable to work, on Medical Leave | 4
Marital Status [Count of Participants; unit: Participants]
  Never Married | 7
  Divorced or Separated | 5
  Widowed | 2
  Presently Married or Living with Partner | 12
Gynecological History [Count of Participants; unit: Participants]
  Perimenopausal | 5
  Naturally Postmenopausal | 18
  Surgically Postmenopausal | 3
Years since last menstrual period (LMP) [Count of Participants; unit: Participants]
  <1 Years | 5
  1-5 Years | 13
  >5 Years | 8
Number of Children [Count of Participants; unit: Participants]
  No Children | 12
  1 to 4 Children | 14
Smoking History [Count of Participants; unit: Participants]
  Current Smoker | 4
  Non-Current Smoker | 22
Baseline BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.4 (6.6)
Provider Status [Count of Participants; unit: Participants]
  Has Doctor/Nurse Providing Regular Care | 25
  Does not have Doctor/Nurse Providing Regular Care | 1

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of Gabapentin
Description: Tolerability of gabapentin was assessed by self-report at the week 1, week 4 and week 7 contacts by asking participants to complete the SAFTEE-SI and CPFQ questionnaires and prompting subjects to report any adverse events at each study visit. Tolerability of gabapentin is defined as the proportion of participants that is able to increase the dose from 300-mg to 600-mg and to remain on the higher dose for the duration of the trial.
Time Frame: Baseline, Week 4 visit, and study completion at 7 weeks
Population: All 26 participants who initiated treatment with gabapentin were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Gabapentin
Number analyzed (Participants) | 26
Participants
  # of subjects who tolerated gabapentin | 22
  # of subjects who did not tolerate gabapentin | 4

2. Primary Outcome: Reason for Non-tolerability and Discontinuation of Gabapentin
Description: Reason why subjects who initiated treatment with gabapentin chose to discontinue before study completion
Time Frame: Baseline, Week 4 Visit, and study completion at 7 weeks
Population: Four subjects initiated treatment with gabapentin but discontinued prior to study completion due to side effects.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Gabapentin
Number analyzed (Participants) | 4
Participants
  Morning sickness and Nausea | 3
  Mild Rash | 1

3. Primary Outcome: Vasomotor Symptoms (VMS) Frequency, Severity, and Bothersomeness During Daytime
Description: Vasomotor symptoms (VMS) were tracked and quantified prospectively using a daily hot flash diary. The hot flash diary was adapted from a 7-day self-report tool for vasomotor symptoms originally developed by the North Central Cancer Treatment Group (NCCTG). The diary asks for the subject to log number of hot flashes during the day and night, severity of hot flashes during day and night, and how bothersome the hot flashes were during day and night. Vasomotor symptoms were also systematically assessed at baseline, week 4, and week 7 using the Hot Flash-Related Daily Interference Scale (HFRDIS), a 10-item self-report questionnaire to determine perceived hot flash interference with quality of life and daily activities.
Time Frame: Baseline, study completion at 7 weeks
Population: Though 20 participants completed the study, the analyzable population includes only the 19 completers who have VMS data for both baseline and the final visit.
Measure: Mean (Full Range); unit: vasomotor symptoms (VMS) per day
Arm/Group | Open-label Gabapentin
Number analyzed (Participants) | 19
vasomotor symptoms (VMS) per day
  mean VMS per day at baseline | 4.1 [0.2 to 8.5]
  mean VMS per day at study completion | 2.2 [0 to 6.7]

4. Primary Outcome: Vasomotor Symptoms (VMS) Frequency, Severity, and Bothersomeness During Nighttime
Description: as for outcome 3
Time Frame: Baseline, study completion at 7 weeks
Population: as for outcome 3
Measure: Mean (Full Range); unit: vasomotor symptoms (VMS) per night
Arm/Group | Open-label Gabapentin
Number analyzed (Participants) | 19
vasomotor symptoms (VMS) per night
  mean VMS per night at baseline | 3.5 [1.5 to 8.0]
  mean VMS per night at study completion | 1.1 [0 to 3.9]

5. Primary Outcome: Severity of Insomnia
Description: Severity of insomnia was measured throughout the study using the Insomnia Severity Index (ISI) .The ISI is a 7-item scale that evaluates the severity of insomnia retrospectively over the past week. The scale is more specific to insomnia symptoms than the Pittsburgh scale (PSQI), which focuses more broadly on overall sleep quality.
  The ISI score ranges from a minimum of 0 to 28. A score of 0-7=no clinically significant insomnia, 8-14=subthreshold insomnia, 5-21=clinical insomnia (moderate severity), 22-28=clinical insomnia (severe), with higher values indicating more severe insomnia.
Time Frame: Baseline, study completion at 7 weeks
Population: Analyzable population includes all 20 completers of the study, since all 20 completers of the study had ISI data at baseline and study completion.
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Open-label Gabapentin
Number analyzed (Participants) | 20
scores on a scale
  mean ISI score at baseline | 15.6 [8 to 24]
  mean ISI score at study completion | 6.0 [0 to 18]

6. Primary Outcome: Sleep Quality and Disturbances Over Past Month
Description: Sleep quality and disturbances during the past month were assessed with the Pittsburgh Sleep Quality Index (PSQI). The PSQI also incorporates daytime functioning into the total score.
  In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Time Frame: Baseline, study completion at 7 weeks
Population: Analyzable population includes all 20 completers of the study, since all 20 completers of the study had PSQI data at baseline and study completion.
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Open-label Gabapentin
Number analyzed (Participants) | 20
scores on a scale
  PSQI total score at baseline | 9.6 [4 to 17]
  PSQI total score at study completion | 4.9 [0 to 12]

7. Other Pre Specified Outcome: Quality of Life-Overall
Description: Quality of life-Overall was assessed with the Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q). The Q-LES-Q is a 16-item self-report questionnaire that assesses enjoyment of and satisfaction with life. The scoring of the Q-LES-Q-SF involves summing only the first 14 items to yield a raw total score. The last two items are not included in the total score but are standalone items. The raw total score ranges from 14 to 70 with higher scores indicating higher quality of life enjoyment and satisfaction.
Time Frame: Baseline, study completion at 7 weeks
Population: Analyzable population includes all 20 completers of the study, since all 20 completers of the study had Q-LES-Q data at baseline and study completion.
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Open-label Gabapentin
Number analyzed (Participants) | 20
scores on a scale
  Q-LES-Q scores at baseline | 60.3 [30 to 80]
  Q-LES-Q scores at study completion | 61.7 [35 to 80]

8. Other Pre Specified Outcome: Quality of Life-Menopause Specific
Description: The Quality of life-Menopause specific is assessed by the Menopause Specific Quality of Life (MENQOL).
  The MENQOL is self-administered and consists of a total of 29 items in a Likert-scale format. Each item assesses the impact of one of four domains of menopausal symptoms, as experienced over the last month: vasomotor (items 1-3), psychosocial (items 4-10), physical (items 11-26), and sexual (items 27-29). Items pertaining to a specific symptom are rated as present or not present, and if present, how bothersome on a zero (not bothersome) to six (extremely bothersome) scale. Means are computed for each subscale by dividing the sum of the domain's items by the number of items within that domain. Non-endorsement of an item is scored a "1" and endorsement a "2," plus the number of the particular rating, so that the possible score on any item ranges from 1-8. Total score also ranges from 1-8.
Time Frame: Baseline, study completion at 7 weeks
Population: Analyzable population includes all 20 completers of the study, since all 20 completers of the study had MENQOL data at baseline and study completion.
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Open-label Gabapentin
Number analyzed (Participants) | 20
scores on a scale
  MENQOL scores at baseline | 3.2 [1 to 5]
  MENQOL scores at study completion | 1.9 [1 to 3.5]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected using the SAFTEE-SI self-report questionnaire at each visit
Arm/Group | Open-label Gabapentin
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 11/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Gabapentin (N=26)
Headaches (Nervous system disorders) | 9
Sweating (Respiratory, thoracic and mediastinal disorders) | 8
Hot flashes (Pregnancy, puerperium and perinatal conditions) | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Feeling tired/fatigue (General disorders) | 6
Feeling drowsy during the day (General disorders) | 8
Problems falling asleep (General disorders) | 4
Weight gain (Metabolism and nutrition disorders) | 4
Stomach/abdominal discomfort (Gastrointestinal disorders) | 4
Gas (Gastrointestinal disorders) | 4
Tension (Psychiatric disorders) | 4
Increased interest in sex (Reproductive system and breast disorders) | 4
Waking up too early (General disorders) | 4
Coughing (Respiratory, thoracic and mediastinal disorders) | 4
Aches, pains in muscles, bones or joints (Musculoskeletal and connective tissue disorders) | 4
Nausea (General disorders) | 3
Mild rash (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
* lack of control group (important given that previous VMS medication trials have indicated modest placebo response rates)
* small sample size
* relatively low rate of completion (6 of 26 subjects who received medication did not reach study endpoint)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No